CLINICAL TRIAL: NCT03173261
Title: Role of Genexpert in Extra Pulmonary Tuberculosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, lamia saad, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PTB
Record Dates: First submitted 2017-05-23; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Extra Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Extrapulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tuberculous pleural effusion (Other): diagnosis of tuberculous pleural effusion and genitourinary tuberculosis by Genexpert by urine and pus and pleural fluid aspirate
  Interventions: Diagnostic Test: Genexpert

INTERVENTIONS:
Diagnostic Test: Genexpert — diagnosis of tuberculous pleural effusion and genitourinary tuberculosis by Genexpert by urine and pus and pleural fluid aspirate

SUMMARY:
Diagnosis of extra pulmonary tuberculosis remains especially challenging since the number of Mycobacterium tuberculosis bacilli present in tissues at sites of disease is often low and clinical specimens from deep-seated organs may be difficult to obtain. Histology is time-consuming to undertake and establishing a diagnosis of tuberculosis with high specificity remains difficult. Tissue microscopy after special staining is often negative and when mycobacteria are seen, it is impossible to distinguish Mycobacterium tuberculosis from non tuberculous mycobacterial disease. Reliance on culture, the mainstay of diagnosis, often leads to considerable delays, compromising patient care and outcomes.

Evidence from 138 studies published before 2008 suggested that nucleic acid amplification technologies could not replace conventional mycobacterial tests (microscopy, culture) for diagnosing pulmonary and, especially, extra pulmonary tuberculosis

DETAILED DESCRIPTION:
Only a few years later, GeneXpert technology has changed this paradigm, with a recent systematic review showing pooled sensitivity of 88% and pooled specificity of 98% for diagnosis of pulmonary tuberculosis, but evidence (as of March 2012) for using Xpert MTB/RIF for diagnosing extra pulmonary tuberculosis is still comparatively weak Globally, there is still a dearth of studies involving the use of Xpert MTB/RIF in extra pulmonary tuberculosis specimens, and few provide definitive answers. This is due mostly to the studies having small sample sizes across a range of various specimen types and differences in pre-processing methodologies and in input volumes and to studies having been conducted in different populations (adults, children, Human immunodeficiency virus infected).

ELIGIBILITY:
Inclusion Criteria:

* All patients with extra pulmonary tuberculosis

Exclusion Criteria:

* Severe co morbid diseases.
* pulmonary tuberculosis
* patients refuse to do genexpert or refusing

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
the percentage of positive patients for extra pulmonary tuberculosis | 10 minutes
  Count of tuberculosis bacilli in the specimen

CONTACTS AND LOCATIONS:
Overall Officials: Raafat Talett, Study Chair — Assiut University; Yaser Ahmed, Study Chair — Assiut University; Ahmed Metwally, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boehme CC, Nabeta P, Hillemann D, Nicol MP, Shenai S, Krapp F, Allen J, Tahirli R, Blakemore R, Rustomjee R, Milovic A, Jones M, O'Brien SM, Persing DH, Ruesch-Gerdes S, Gotuzzo E, Rodrigues C, Alland D, Perkins MD. Rapid molecular detection of tuberculosis and rifampin resistance. N Engl J Med. 2010 Sep 9;363(11):1005-15. doi: 10.1056/NEJMoa0907847. Epub 2010 Sep 1. PMID 20825313
- [Result] Lawn SD, Zumla AI. Tuberculosis. Lancet. 2011 Jul 2;378(9785):57-72. doi: 10.1016/S0140-6736(10)62173-3. Epub 2011 Mar 21. PMID 21420161